CLINICAL TRIAL: NCT00117611
Title: Effects of Anti-IgE Antibody Omalizumab (Xolair) on Patients With Chronic Sinusitis and a Positive Allergen Test
Brief Title: Xolair in Patients With Chronic Sinusitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Genentech, Inc. (Industry); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13916A; Q2347s
Record Dates: First submitted 2005-06-30; First posted 2005-07-07 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Sinusitis
Keywords: chronic sinusitis
MeSH Terms: conditions — Sinusitis | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Xolair administered subcutaneously, once or twice monthly (dose dependent on subject weight and serum IgE level)
  Interventions: Drug: Anti-IgE antibody omalizumab or placebo
- 2 (Placebo Comparator): placebo administered subcutaneously once or twice monthly
  Interventions: Drug: Anti-IgE antibody omalizumab or placebo

INTERVENTIONS:
Drug: Anti-IgE antibody omalizumab or placebo — given subcutaneously oce or twice monthly depending on dose
  Other Names: Xolair or placebo

SUMMARY:
The purpose of this study is to determine if treatment with the anti-IgE antibody, Xolair (omalizumab), will improve objective and subjective evidence of chronic sinusitis.

DETAILED DESCRIPTION:
At its most basic level, sinusitis is defined as an inflammation of the lining membrane of the paranasal sinuses. Sinusitis affects all age groups, including 17% of people above the age of 65 years. On the basis of national population surveys and insurance-reimbursement claims, sinusitis is one of the most common health problems in the U.S. Thus, each year, billions of dollars are spent on direct medical costs for the treatment of this enigmatic illness.

Despite the enormous cost of the problem, there are no definite studies of treatment and management. There are some data indicating that intranasal steroids are effective, and recently Nasonex was approved for the treatment of nasal polyps. All other treatments are empirically based.

There is evidence that IgE antibodies play a role in chronic sinusitis. The investigators have shown that total IgE levels correlate with the severity of sinusitis, as assessed by CT scan. Staphylococcus enterotoxins cause local increases in total IgE in over 50% of nasal polyp patients. Allergies occur more frequently in patients with chronic sinusitis than in the general population. Elevations in total IgE have been shown to occur in patients with allergic fungal sinusitis and the levels of total IgE decrease with successful treatment. Thus, the investigators speculate that IgE contributes significantly to the pathogenesis of chronic sinusitis.

The purpose of this study is to determine if treatment with the anti-IgE antibody, Xolair, will improve objective and subjective evidence of chronic sinusitis.

ELIGIBILITY:
Inclusion Criteria:

* Chronic sinusitis, as defined by symptoms for greater than 12 weeks, despite treatment
* Paranasal sinus CT scan showing evidence of chronic sinusitis
* Positive skin or RAST test to an inhalant allergen
* Serum total IgE between 30 and 700 International Units/ml
* Body weight less than 150 kg
* Impaired quality of life, as measured by the Rhinosinusitis Disability Index (RSDI)

Exclusion Criteria:

* Women of childbearing potential not using a contraception method(s) (birth control pills, Depo Provera, double barrier) as well as women who are breastfeeding
* Known sensitivity to Xolair
* Patients with severe medical condition(s) that, in the opinion of the investigator, prohibits participation in the study (heart, lung, kidney, neurological, oncologic or liver disease)
* Use of any other investigational agent in the last 30 days
* No measurable disability on the RSDI
* Immunocompromised patients or patients with ciliary disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2005-07; Primary Completion 2007-05 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Mucosal thickness on CT scan | after 6 months of treatment

SECONDARY OUTCOMES:
Rhinosinusitis Disability Index (RSDI)recorded monthly | 6 months
A specific quality of life (QOL) measure, Sino-Nasal Outcome Test (SNOT 20)recorded monthly | 6 months
A general health QOL measure (SF-36) | 6 months
The number of sinusitis exacerbations requiring additional treatment | 6 months
Nasal peak inspiratory flow | 6 months
Symptoms of nasal discharge, nasal obstruction, facial pain and altered smell | 6 months
Nasal lavage eosinophils | 6 months
Nasal endoscopy score | 6 months
The University of Pennsylvania Smell Identification Test (UPSIT) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Naclerio, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Benninger MS, Senior BA. The development of the Rhinosinusitis Disability Index. Arch Otolaryngol Head Neck Surg. 1997 Nov;123(11):1175-9. doi: 10.1001/archotol.1997.01900110025004. PMID 9366696
- [Background] Piccirillo JF, Merritt MG Jr, Richards ML. Psychometric and clinimetric validity of the 20-Item Sino-Nasal Outcome Test (SNOT-20). Otolaryngol Head Neck Surg. 2002 Jan;126(1):41-7. doi: 10.1067/mhn.2002.121022. PMID 11821764
- [Background] Busse W, Corren J, Lanier BQ, McAlary M, Fowler-Taylor A, Cioppa GD, van As A, Gupta N. Omalizumab, anti-IgE recombinant humanized monoclonal antibody, for the treatment of severe allergic asthma. J Allergy Clin Immunol. 2001 Aug;108(2):184-90. doi: 10.1067/mai.2001.117880. PMID 11496232
- [Background] Soler M, Matz J, Townley R, Buhl R, O'Brien J, Fox H, Thirlwell J, Gupta N, Della Cioppa G. The anti-IgE antibody omalizumab reduces exacerbations and steroid requirement in allergic asthmatics. Eur Respir J. 2001 Aug;18(2):254-61. doi: 10.1183/09031936.01.00092101. PMID 11529281
- [Background] Calhoun KH, Waggenspack GA, Simpson CB, Hokanson JA, Bailey BJ. CT evaluation of the paranasal sinuses in symptomatic and asymptomatic populations. Otolaryngol Head Neck Surg. 1991 Apr;104(4):480-3. doi: 10.1177/019459989110400409. PMID 1903859
- [Background] Iwabuchi Y, Hanamure Y, Ueno K, Fukuda K, Furuta S. Clinical significance of asymptomatic sinus abnormalities on magnetic resonance imaging. Arch Otolaryngol Head Neck Surg. 1997 Jun;123(6):602-4. doi: 10.1001/archotol.1997.01900060044007. PMID 9193220
- [Background] McCaig LF, Hughes JM. Trends in antimicrobial drug prescribing among office-based physicians in the United States. JAMA. 1995 Jan 18;273(3):214-9. PMID 7807660
- [Background] Kaliner MA, Osguthorpe JD, Fireman P, Anon J, Georgitis J, Davis ML, Naclerio R, Kennedy D. Sinusitis: bench to bedside. Current findings, future directions. Otolaryngol Head Neck Surg. 1997 Jun;116(6 Pt 2):S1-20. PMID 9212028
- [Background] Hamilos DL. Chronic sinusitis. J Allergy Clin Immunol. 2000 Aug;106(2):213-27. doi: 10.1067/mai.2000.109269. PMID 10932063
- [Background] Iwens P, Clement PA. Sinusitis in allergic patients. Rhinology. 1994 Jun;32(2):65-7. PMID 7939142
- [Background] Binder E, Holopainen E, Malmberg H, Salo OP. Clinical findings in patients with allergic rhinitis. Rhinology. 1984 Dec;22(4):255-60. PMID 6522975
- [Background] Rachelefsky GS, Goldberg M, Katz RM, Boris G, Gyepes MT, Shapiro MJ, Mickey MR, Finegold SM, Siegel SC. Sinus disease in children with respiratory allergy. J Allergy Clin Immunol. 1978 May;61(5):310-4. doi: 10.1016/0091-6749(78)90052-0. No abstract available. PMID 641266
- [Background] Holzmann D, Willi U, Nadal D. Allergic rhinitis as a risk factor for orbital complication of acute rhinosinusitis in children. Am J Rhinol. 2001 Nov-Dec;15(6):387-90. PMID 11777246
- [Background] Chen CF, Wu KG, Hsu MC, Tang RB. Prevalence and relationship between allergic diseases and infectious diseases. J Microbiol Immunol Infect. 2001 Mar;34(1):57-62. PMID 11321129
- [Background] VAN DISHOECK HA, FRANSSEN MG. The incidence and correlation of allergy and chronic maxillary sinusitis. Pract Otorhinolaryngol (Basel). 1957 Nov;19(6):502-6. doi: 10.1159/000274105. No abstract available. PMID 13494297
- [Background] Friedman WH. Surgery for chronic hyperplastic rhinosinusitis. Laryngoscope. 1975 Dec;85(12 pt 1):1999-2011. doi: 10.1288/00005537-197512000-00005. PMID 1202305
- [Background] Enberg RN. Perennial nonallergic rhinitis: a retrospective review. Ann Allergy. 1989 Dec;63(6 Pt 1):513-6. PMID 2480728
- [Background] Conner BL, Roach ES, Laster W, Georgitis JW. Magnetic resonance imaging of the paranasal sinuses: frequency and type of abnormalities. Ann Allergy. 1989 May;62(5):457-60. PMID 2719356
- [Background] Settipane GA, Chafee FH. Nasal polyps in asthma and rhinitis. A review of 6,037 patients. J Allergy Clin Immunol. 1977 Jan;59(1):17-21. doi: 10.1016/0091-6749(77)90171-3. PMID 833373
- [Background] Holmberg K, Juliusson S, Balder B, Smith DL, Richards DH, Karlsson G. Fluticasone propionate aqueous nasal spray in the treatment of nasal polyposis. Ann Allergy Asthma Immunol. 1997 Mar;78(3):270-6. doi: 10.1016/s1081-1206(10)63180-8. PMID 9087151
- [Background] Lund VJ, Flood J, Sykes AP, Richards DH. Effect of fluticasone in severe polyposis. Arch Otolaryngol Head Neck Surg. 1998 May;124(5):513-8. doi: 10.1001/archotol.124.5.513. PMID 9604976
- [Background] Karlsson G, Holmberg K. Does allergic rhinitis predispose to sinusitis? Acta Otolaryngol Suppl. 1994;515:26-8; discussion 29. doi: 10.3109/00016489409124319. PMID 8067239
- [Background] Kingdom TT, Lee KC, FitzSimmons SC, Cropp GJ. Clinical characteristics and genotype analysis of patients with cystic fibrosis and nasal polyposis requiring surgery. Arch Otolaryngol Head Neck Surg. 1996 Nov;122(11):1209-13. doi: 10.1001/archotol.1996.01890230055011. PMID 8906056
- [Derived] Pinto JM, Mehta N, DiTineo M, Wang J, Baroody FM, Naclerio RM. A randomized, double-blind, placebo-controlled trial of anti-IgE for chronic rhinosinusitis. Rhinology. 2010 Sep;48(3):318-24. doi: 10.4193/Rhino09.144. PMID 21038023